CLINICAL TRIAL: NCT04202510
Title: Pressure Reduction and Medication Use Following Different Minimally Invasive Glaucoma Surgery Procedures, Prospective Randomized Clinical Trial of Efficacy
Brief Title: IOP and Medication Reduction in MIGS Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and the decrease in surgical cases, sufficient patients were not available.
Sponsor: Wills Eye (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Daniel Lee, MD, Principle Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #19-869
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Open Angle Glaucoma; Primary Open Angle Glaucoma; Pigmentary Glaucoma; Pseudoexfoliation Glaucoma in Both Eyes
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- iStent (Active Comparator): iStent Trabecular Bypass Device (to lower intraocular pressure) combined with Phacoemulsification (to remove cataract and insert intraocular lens) Eye Surgery
  Interventions: Procedure: Glaucoma and Cataract Surgery
- iStent Inject (Active Comparator): iStent Inject Trabecular Bypass Device (to lower intraocular pressure) combined with Phacoemulsification (to remove cataract and insert intraocular lens) Eye Surgery
  Interventions: Procedure: Glaucoma and Cataract Surgery
- Hydrus (Active Comparator): Hydrus Trabecular Bypass Device (to lower intraocular pressure) combined with Phacoemulsification (to remove cataract and insert intraocular lens) Eye Surgery
  Interventions: Procedure: Glaucoma and Cataract Surgery

INTERVENTIONS:
Procedure: Glaucoma and Cataract Surgery — Patients requiring combined cataract and glaucoma surgery will be randomized to either iStent, iStent Inject or Hydrus (to lower intraocular pressure) combined with Phacoemulsification (to remove cataract and insert intraocular lens) Eye Surgery

SUMMARY:
The primary objective of this research is to compare the efficacy of trabecular minimally invasive glaucoma surgery (MIGS) devices (iStent vs iStent Inject vs Hydrus) for intra ocular pressure (IOP) and anti-glaucoma medication reduction in open angle glaucoma.

DETAILED DESCRIPTION:
Study Design Prospective Randomized Clinical Trial (Parallel Group Study)

Patients who fit inclusion criteria will be randomly assigned to one of the 3 parallel groups (one of the study surgical interventions combined with phacoemulsification) in the following order:

1. 1st Generation iStent, Trabecular Micro-Bypass Device (Glaukos Inc, San Clemente, CA).
2. 2nd Generation iStent, Trabecular Micro-Bypass Device (Glaukos Inc, San Clemente, CA).
3. Hydrus Microstent (Ivantis Inc, Irvine, CA). Blocked randomization will be used in 1:1:1 ratio to provide balanced study groups. Allocation will be performed using a random number table.

Preoperative Evaluation of : Visual acuity, Slit lamp examination, IOP, Gonioscopy, Fundus Examination, Central corneal thickness (CCT), Endothelial Cell Count (ECC), Visual field, Retinal Nerve Fiber layer (RNFL) thickness by Optical Coherence Tomography (OCT) and Number and type of preoperative antiglaucoma medications.

Patients will be followed postoperatively at Day 1, Week 1, Months 1, 3, 6 and 12.

Medication Washout will be done at baseline, Months 6 and 12 to evaluate non-medicated IOP.

The duration of washout will be:

4 Weeks for Prostaglandin Analogues (PGA) and Beta Blockers (BB). 2 Weeks for Carbonic Anhydrase Inhibitors (CAI) and Alpha Agonists (AA).

The IOP measurements in the wash out visits:

will be performed according to 2-operator method to provide masking as described in Ocular Hypertension Treatment Study (OHTS) and Glaucoma World Association Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult male or female aged 40 years or more. 2. Patients able and willing to provide informed consent. 3. Patients having Visually Significant Age Related Cataract with Mild to Moderate Open Angle Glaucoma (OAG) on topical anti-glaucoma medication with or without previous Selective Laser Trabeculoplasty (SLT) ), including:

  1. Primary open angle glaucoma (POAG).
  2. Pigmentary glaucoma.
  3. Pseudoexfoliative glaucoma. 4. Patients should be candidate for safe mediaction wash out in the opinion of the investigator.

     * The diagnosis of glaucoma is confirmd by optic nerve examination and the characteristic visual field defects on automated perimetry according to the American Academy of Ophthalmology (AAO) Definition and Criteria.
     * The severity of glaucoma is classified using the Hodapp Parrish Anderson Visual Field Criteria depending on the Mean Deviation (MD):

       1. Mild: MD no worse than -6 dB.
       2. Moderate: MD worse than -6 but no worse than -12 dB.
       3. Severe: MD worse than -12 dB.

Exclusion Criteria:

1. Glaucoma types rather than open angle glaucoma types mentioned in the inclusion criteria (Primary, Pigmentary and Pseudoexfoliation Glaucomas).
2. Any prior glaucoma, corneal or vitreoretinal surgery.
3. Evidence of concomitant retinal, optic nerve, or neurological diseases affecting the visual field.
4. Abnormal angle anatomy.
5. Prior Argon Laser Trabeculoplasty (ALT), Laser Iridotomy or Iridoplasty.
6. Any systemic condition or medications affectiong IOP.
7. Corneal opacity, corneal dystrophy or central corneal thickness (CCT) less than 480 or more than 620 microns.
8. Exclusion from medications wash out according to the opinion of the investigator Or if any of the following is observed at any time point of the study:

   1. Visual Field: Mean deviation worse than -12 dB.
   2. Intraocular pressure: a treated IOP of greater than 24 mmHg.
   3. Medications: using more than three medications.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 1 hour examination at Baseline, Day 1, Week 1, Months 1, 3, 6 and 12
  Reduction of IOP after eye surgery measured in millimeters of mercury (mmHg)

SECONDARY OUTCOMES:
Visual Acuity | 1 hour examination at Baseline, Day 1, Week 1, Months 1, 3, 6 and 12
  Change in visual acuity after eye surgery measured in minimal angle of resolution (logMAR).
Central Corneal Thickness (CCT) | 1 hour examination at Baseline, Months 3, 6 and 12
  Change in CCT after eye surgery measured in microns using pachymeter.
Endothelial Cell Count | 1 hour examination at Baseline, Months 3, 6 and 12
  Change in endothelial cell count after eye surgery measured in number of cells by millimeter square using specular microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No